CLINICAL TRIAL: NCT02059174
Title: A Single Dose Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-1293 and to Compare Its Pharmacologic Properties to Those of Another Basal Insulin in Subjects With Type I Diabetes
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-1293 Compared With a Basal Insulin in Participants With Type 1 Diabetes (MK-1293-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1293-005; 2012-005656-41 (EudraCT Number)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — MK-1293; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-1293 / EU-Lantus™ / MK-1293 / EU-Lantus™ (Experimental): MK-1293 or EU-Lantus™ 0.4 units/kg administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design with a minimum of 7 days between each treatment period
  Interventions: Drug: MK-1293; Drug: EU-Lantus™; Drug: Novolog™
- EU-Lantus™ / MK-1293 / EU-Lantus™ / MK-1293 (Experimental): MK-1293 or EU-Lantus™ 0.4 units/kg administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design with a minimum of 7 days between each treatment period
  Interventions: Drug: MK-1293; Drug: EU-Lantus™; Drug: Novolog™

INTERVENTIONS:
Drug: MK-1293 — MK-1293 0.4 units/kg administered subcutaneously
Drug: EU-Lantus™ — EU-Lantus™ 0.4 units/kg administered subcutaneously
Drug: Novolog™ — Participants will receive an intravenous infusion of insulin aspart (Novolog™ or other rapid-acting insulin analog) for several hours prior to MK-1293 or EU-Lantus™ dosing in each dosing period to meet basal insulin requirements

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics, and pharmacodynamics of MK-1293 compared with a basal insulin (EU-Lantus™) in participants with Type 1 Diabetes. The primary hypotheses are that the duration of action, pharmacodynamic profile, and pharmacokinetic profile of MK-1293 and the comparator basal insulin are similar.

ELIGIBILITY:
Inclusion Criteria:

* Has type 1 diabetes mellitus diagnosed at least 12 months before screening
* Subject to investigator discretion, is on a stable dose of insulin for at least 2 weeks before screening
* Has a total daily insulin dose <=1.2 units/kg
* Has a screening hemoglobin A1c <9.5%
* Has a body mass index >18.0 and <=30.0 kg/m^2
* Has a weight >=50 kg
* Female participant of reproductive potential has a serum beta-human chorionic gonadotropin level consistent with the nongravid state and agrees to use (and/or have her partner use) 2 acceptable methods of birth control until 2 weeks after the last dose of study drug
* Postmenopausal female participant is without menses for >=1 year
* Surgically sterile female participant status is post hysterectomy, oophorectomy, or tubal ligation
* Has not used nicotine or nicotine-containing products for at least 3 months before study start or smokes less than 10 cigarettes per day and is willing to abstain during the trial

Exclusion Criteria:

* Has a history of clinically significant gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or disease
* Has a history of clinically significant endocrine abnormalities or diseases except type 1 diabetes mellitus
* Has had any severe hypoglycemic episodes associated with hypoglycemic seizures, comas, or unconsciousness within the past 3 months
* Has a history of diabetic ketoacidosis within the past 6 months
* Has a history of significant multiple or severe allergies, anaphylactic reaction, or significant intolerability to drugs or food
* Has a history of hypersensitivity to pharmacologic insulins
* Is positive for hepatitis B surface antigen, hepatitis C, or Human Immunodeficiency Virus
* Has had major surgery or donated or lost 1 unit of blood within 4 weeks before screening
* Unable to refrain from use of any medication or herbal remedy from 2 weeks prior to the first dose of study drug to until the posttrial visit. Some medications are permitted and may be discussed with the investigators
* Vaccination within 12 weeks of start of study participation
* Consumes >3 glasses of alcoholic beverages per day. Participants consuming 4 glasses of alcoholic beverages may be enrolled at the discretion of the investigator.
* Consumes >6 servings of caffeinated beverages per day
* Is a regular user of any illicit drugs or has a history of drug abuse (including alcohol) within approximately 1 year
* Is on a carbohydrate-restricted diet (<100 grams carbohydrate per day); participants who are on a carbohydrate-restricted diet may be included if they agree to a diet consisting of >=100 grams of carbohydrate daily throughout the study
* Has a personal or family history of hypercoagulability or thromboembolic disease
* Has used systemic glucocorticoids within 3 months of screening or anticipates treatment with systemic glucocorticoids during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2015-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Crutchlow MF, Palcza JS, Mostoller KM, Mahon CD, Barbour AM, Marcos MC, Xu Y, Watkins E, Morrow L, Hompesch M. Single-dose euglycaemic clamp studies demonstrating pharmacokinetic and pharmacodynamic similarity between MK-1293 insulin glargine and originator insulin glargine (Lantus) in subjects with type 1 diabetes and healthy subjects. Diabetes Obes Metab. 2018 Feb;20(2):400-408. doi: 10.1111/dom.13084. Epub 2017 Sep 26. PMID 28817223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants with Type I diabetes mellitus between the ages of 18 and 65 years (inclusive) were enrolled in this trial in 1 clinical site in the United States.
Period: Period 1
Arm/Group | MK-1293 / EU-Lantus™ / MK-1293 / EU-Lantus™ | EU-Lantus™ / MK-1293 / EU-Lantus™ / MK-1293
Started | 37 | 39
Completed | 37 | 37
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 2
Arm/Group | MK-1293 / EU-Lantus™ / MK-1293 / EU-Lantus™ | EU-Lantus™ / MK-1293 / EU-Lantus™ / MK-1293
Started | 37 | 37
Completed | 36 | 35
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 1 | 0
Period: Period 3
Arm/Group | MK-1293 / EU-Lantus™ / MK-1293 / EU-Lantus™ | EU-Lantus™ / MK-1293 / EU-Lantus™ / MK-1293
Started | 36 | 35
Completed | 35 | 35
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Period 4
Arm/Group | MK-1293 / EU-Lantus™ / MK-1293 / EU-Lantus™ | EU-Lantus™ / MK-1293 / EU-Lantus™ / MK-1293
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: MK-1293 or EU-Lantus™ 0.4 units/kg administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design with a minimum of 7 days between each treatment period
Arm/Group | All Participants
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Comparison of MK-1293 and EU-Approved Lantus Duration of Pharmacodynamic Action During a 30-Hour Euglycemic Clamp Study
Description: Duration of Action (DOA) is defined as the length of time from dosing to End of Action. End of Action is defined as the time point at which plasma glucose has been above 150 mg/dL for 30 minutes and no glucose has been infused for 30 minutes. Median and max below are reported for the length of clamp duration (i.e. 30 hours).
Time Frame: Up to 30 hours postdose
Population: The Per-Protocol population consists of 75 participants, including the 70 with complete data across all 4 treatment periods and 5 participants with partial data. One participant was not included in the PP population due to a medical issue. All available data from 5 of the participants who discontinued the study were included in the analyses.
Measure: Median (Full Range); unit: Hours
Groups:
- MK-1293: MK-1293 0.4 units/kg administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design with a minimum of 7 days between each treatment period
- EU-Lantus™: EU-Lantus™ 0.4 units/kg administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design with a minimum of 7 days between each treatment period
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 75
Hours | 30 [0 to 30] | 30 [11.93 to 30]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Because numerous participants did not achieve End of Action within the 30-hour clamp timeframe, the pre-specified hypothesis of similarity with regard to mean DOA could not be tested and a survival analysis approach was undertaken. The hazard rate is a measure of the instantaneous risk of reaching End of Action at time t given End of Action has not been met up until time t, with the hazard ratio being an estimate of the relative difference in hazard rates between treatments; Test type: Non-Inferiority or Equivalence — A frailty model was used with effects for treatment, period and sequence and a random effect for participant. A value of 1.00 for the hazard ratio corresponds to no difference between treatments; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.72 to 1.59] — ratio (MK-1293 / EU-Approved Lantus)

2. Primary Outcome: PD: Area Under the Glucose Infusion Rate Versus Time Curve Over 24 Hours After Dosing (GIR-AUC0-24hr)
Description: The area under the glucose infusion rate curve from hours 0 to 24 after injection (AUC[GIR{0-24}]) for participants who received either MK-1293 or EU-Lantus™ administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design was measured from blood samples obtained during a euglycemic clamp procedure.
Time Frame: Up to 24 hours postdose
Population: The Per-Protocol population included 70 participants with complete data and 5 participants with partial data. One participant was not included in the PP population due to a medical issue. Data from 5 discontinued participants were included in the analyses; data from 1 participant was not (incomplete clamp data, only out to 18.5 hours).
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 74
mg/kg | 1470.07 [1256.52 to 1683.63] | 1554.53 [1334.03 to 1775.04]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — Similarity criteria calculated via Fieller's Theorem was 95% confidence interval for arithmetic mean ratio (MK-1293/EU-Lantus™) falls between 0.80-1.25; Ratio of Arithmetic Means = 0.95, 95% CI 2-sided [0.88 to 1.01] — Ratio (MK-1293 / EU-Approved Lantus)

3. Primary Outcome: PD: Area Under the Glucose Infusion Rate Versus Time Curve Over the First 12 Hours After Dosing (GIR-AUC0-12hr)
Description: The area under the glucose infusion rate curve from hours 0 to 12 after injection (AUC[GIR{0-12}]) for participants who received either MK-1293 or EU-Lantus™ administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design was measured from blood samples obtained during a euglycemic clamp procedure.
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 75
mg/kg | 659.38 [557.84 to 760.92] | 736.31 [625.22 to 847.41]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of Arithmetic Means = 0.90, 95% CI 2-sided [0.81 to 0.99] — Ratio (MK-1293 / EU-Approved Lantus)

4. Primary Outcome: PD: Area Under the Glucose Infusion Rate Versus Time Curve Over the Second 12 Hours After Dosing (GIR-AUC12-24hr)
Description: The area under the glucose infusion rate curve from hours 12 to 24 after injection (AUC[GIR{12-24}]) for participants who received either MK-1293 or Lantus™ administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design was measured from blood samples obtained during a euglycemic clamp procedure.
Time Frame: From 12 to 24 hours postdose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 74
mg/kg | 811.43 [689.89 to 932.98] | 818.20 [700.40 to 936.01]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of Arithmetic Means = 0.99, 95% CI 2-sided [0.92 to 1.06] — Ratio (MK-1293 / EU-Approved Lantus)

5. Primary Outcome: PD: Maximum Glucose Infusion Rate (GIRmax)
Description: Maximum glucose infusion rate (GIR[max]) based on smoothed data for participants who received either MK-1293 or EU-Lantus™ administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design was measured from blood samples obtained during a euglycemic clamp procedure.
Time Frame: Up to 30 hours postdose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 74
mg/kg/min | 2.34 [2.11 to 2.57] | 2.43 [2.18 to 2.68]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of Arithmetic Means = 0.96, 95% CI 2-sided [0.91 to 1.02] — Ratio (MK-1293 / EU-Approved Lantus)

6. Primary Outcome: M1 Glargine Metabolite Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve (AUC0-24)
Description: M1 glargine is the dominant circulating glargine-derived insulin metabolite after subcutaneous injection and it is pharmacologically active. AUC0-24 is a measure of the total amount of drug in the plasma from the dose to Hour 24. Analysis was performed on log scale with results back transformed to the original scale
Time Frame: Up to 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg∙hr/mL
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 75
pg∙hr/mL | 6530 [5967 to 7145] | 6763 [6162 to 7423]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — Similarity criteria was 90% confidence interval for geometric mean ratio (MK-1293/EU-Lantus™) falls between 0.80-1.25; Geometric Mean Ratio = 0.97, 90% CI 2-sided [0.91 to 1.02] — Ratio (MK-1293 / EU-Approved Lantus)

7. Primary Outcome: M1 Glargine Metabolite PK: Maximum Plasma Concentration (Cmax)
Description: M1 glargine is the dominant circulating glargine-derived insulin metabolite after subcutaneous injection and it is pharmacologically active. Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Analysis was performed on log scale with results back transformed to original scale.
Time Frame: Up to 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 75
pg/mL | 372 [339 to 408] | 382 [350 to 416]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — Similarity criteria was 90% confidence interval for geometric mean ratio (MK-1293/EU-Lantus™) falls between 0.80-1.25; Geometric Mean Ratio = 0.97, 90% CI 2-sided [0.93 to 1.03] — Ratio (MK-1293 / EU-Approved Lantus)

8. Secondary Outcome: M1 Glargine Metabolite PK: Area Under the Plasma Concentration Versus Time Curve Over the First 12 Hours After Dosing (AUC0-12)
Description: M1 glargine is the dominant circulating glargine-derived insulin metabolite after subcutaneous injection and it is pharmacologically active. AUC0-12 is a measure of the total amount of drug in the plasma from the dose to Hour 12. Analysis was performed on log scale with results back transformed to original scale.
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg∙hr/mL
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 75
pg∙hr/mL | 2981 [2714 to 3274] | 3251 [2968 to 3562]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — Similarity criteria was 90% confidence interval for geometric mean ratio (MK-1293/EU-Lantus™) falls between 0.80-1.25; Geometric Mean Ratio = 0.92, 90% CI 2-sided [0.86 to 0.97] — Ratio (MK-1293 / EU-Approved Lantus)

9. Secondary Outcome: M1 Glargine Metabolite PK: Area Under the Plasma Concentration Versus Time Curve Over the Second 12 Hours After Dosing (AUC12-24)
Description: M1 glargine is the dominant circulating glargine-derived insulin metabolite after subcutaneous injection and it is pharmacologically active. AUC12-24 is a measure of the total amount of drug in the plasma from Hour 12 to Hour 24. Analysis was performed on log scale with results back transformed to original scale.
Time Frame: From 12 to 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg∙hr/mL
Arm/Group | MK-1293 | EU-Lantus™
Number analyzed (Participants) | 74 | 75
pg∙hr/mL | 3510 [3205 to 3845] | 3522 [3228 to 3844]
Statistical Analysis 1: Comparison: MK-1293 vs EU-Lantus™; Test type: Non-Inferiority or Equivalence — Similarity criteria was 90% confidence interval for geometric mean ratio (MK-1293/EU-Lantus™) falls between 0.80-1.25; Geometric Mean Ratio = 1.00, 90% CI 2-sided [0.95 to 1.04] — Ratio (MK-1293 / EU-Approved Lantus)

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug (Up to 7 weeks)
Description: All Subjects as Treated population included all participants who received at least one dose of an investigational drug. Two participants discontinued after Period 1 (EU-Lantus) so did not cross-over to MK-1293.
Groups:
- MK-1293 0.4 Units/kg SC: MK-1293 0.4 units/kg administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design with a minimum of 7 days between treatment periods
- EU-Lantus™ 0.4 Units.kg SC: EU-Lantus™ 0.4 units/kg administered subcutaneously on Day 1 in 2 out of 4 study periods in a replicate crossover design with a minimum of 7 days between treatment periods
Arm/Group | MK-1293 0.4 Units/kg SC | EU-Lantus™ 0.4 Units.kg SC
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76
Other Adverse Events (participants affected / at risk) | 60/74 | 56/76
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1293 0.4 Units/kg SC (N=74) | EU-Lantus™ 0.4 Units.kg SC (N=76)
Injection site haemorrhage (General disorders) | 3 (3) | 4 (4)
Vessel puncture site haemorrhage (General disorders) | 6 (6) | 5 (9)
Vessel puncture site pain (General disorders) | 1 (1) | 4 (4)
Vessel puncture site reaction (General disorders) | 6 (6) | 6 (6)
Skin abrasion (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 55 (120) | 50 (111)
Headache (Nervous system disorders) | 3 (3) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.